CLINICAL TRIAL: NCT00164008
Title: Comparison Between Pamidronate and Zoledronic Acid for the Treatment of Heart and Lung Transplant Related Osteopaenia and Osteoporosis
Brief Title: Comparison of Pamidronate With Zoledronic Acid for Transplant Related Bone Loss Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101/02
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Osteopenia; Complications of Heart-lung Transplant; Other Complications of Lung Transplant
MeSH Terms: conditions — Bone Diseases, Metabolic

INTERVENTIONS:
Drug: zoledronic acid vs pamidronate

SUMMARY:
The purpose of this trial is to see whether zoledronic acid is better than pamidronate to treat low bone density in heart and lung transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* reduced bone density as indicated by a bone density T score <-1.in either the lumbar spine or femoral neck
* have undergone or are on the waiting list for heart or lung transplantation
* are receiving adequate calcium and vitamin D therapy
* have provided written informed consent prior to participation in the trial

Exclusion Criteria:

* untreated hypogonadism, hypothyroidism or hyperthyroidism
* acute or major organ rejection or intercurrent illness
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of lumbar spine at 12 months as measured by DEXA.

SECONDARY OUTCOMES:
Bone mineral density of femoral neck at 12 months as measured by DEXA.

CONTACTS AND LOCATIONS:
Overall Officials: Duncan J Topliss, MD, Principal Investigator — The Alfred